CLINICAL TRIAL: NCT06407050
Title: Effect of the Physical Inactivity Durations During the Day on Postprandial Lipid Metabolism the Morning After Exercise
Brief Title: Duration of Physical Inactivity and Postprandial Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00005669
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-hr trial (Experimental): Participants will go through a day of routine step counts and sleep hour monitor, 2 days of being physical active by taking ambulatory steps, 4 hours of physical inactivity intervention, and moderate intensity cycling, and 1 high fat tolerance test.
  Interventions: Behavioral: 4 hours of physical inactivity
- 8-hr Trial (Experimental): Participants will go through a day of routine step counts and sleep hour monitor, 2 days of being physical active by taking ambulatory steps, 8 hours of physical inactivity intervention, and moderate intensity cycling, and 1 high fat tolerance test.
  Interventions: Behavioral: 8 hours of physical inactivity
- 12-hr Trial (Experimental): Participants will go through a day of routine step counts and sleep hour monitor, 2 days of being physical active by taking ambulatory steps, 12 hours of physical inactivity intervention, and moderate intensity cycling, and 1 high fat tolerance test.
  Interventions: Behavioral: 12 hours of physical inactivity

INTERVENTIONS:
Behavioral: 4 hours of physical inactivity — A pedometer will be worn by participants during the whole trial. Steps will be monitored. Participants will be required to reach 8,500 steps per day for the first 2 days. On the third day participants need to take 600 steps hourly for 8 hours from 7 am to 3 pm and another 2,000 steps between 3:40 pm to 4 pm. Participant will then stay inactive from 4 pm to 8 pm and do a cycling for one hour in the lab. During the inactivity period, participants will remain seated and steps are only allowed for food, water, and bathroom use. A 3 day food log will be given to participants to log in their diet. Participant will be asks to mimic the diet between trials. A Fitbit will be worn by participants to record the sleep hours during the trial.
  Arms: 4-hr trial
Behavioral: 8 hours of physical inactivity — A pedometer will be worn by participants during the whole trial. Steps will be monitored. Participants will be required to reach 8,500 steps per day for the first 2 days. On the third day participants need to take 600 steps hourly for 4 hours from 7 am to 11 am and then 2,000 steps between 11:40 am to 12 pm. During the inactivity period, participants will remain seated and steps are only allowed for food, water, and bathroom use. Participant will then stay inactive from 12 pm to 8 pm and do a cycling for one hour in the lab. A 3 day food log will be given to participants to log in their diet. Participant will be asks to mimic the diet between trials. A Fitbit will be worn by participants to record the sleep hours during the trial.
  Arms: 8-hr Trial
Behavioral: 12 hours of physical inactivity — A pedometer will be worn by participants during the whole trial. Steps will be monitored. Participants will be required to reach 8,500 steps per day for the first 2 days. On the third day, participant will take 2,000 steps between 7:40 am to 8 am and then stay inactive from 8 am to 8 pm. During the inactivity period, participants will remain seated and steps are only allowed for food, water, and bathroom use. Right after the inactivity intervention, participant will do a 1-hr cycling in lab. A 3 day food log will be given to participants to log in their diet. Participant will be asks to mimic the diet between trials. A Fitbit will be worn by participants to record the sleep hours during the trial.
  Arms: 12-hr Trial

SUMMARY:
The purpose of the study is to investigate the effect of different periods of physical inactivity on postprandial lipid metabolism in the morning after exercise by measuring plasma triglyceride levels and fat oxidation (burning). The study is a crossover intervention with all healthy participants performing three trials varying in length of physical inactive (4 hours, 8 hours, and 12 hours). All trials include a physical activity control phase (>8,500 steps/24hr), a physical inactive phase, a moderate intensity cycling session, and a high-fat tolerance test.

DETAILED DESCRIPTION:
This study investigates the effect of the length of physical inactivity during the day on postprandial lipid metabolism the following morning after exercise. Three intervention trials differentiate with different periods of physical inactivity (4 hours, 8 hours, and 12 hours) will be involved for this purpose. The study aims to determine how long a period of physical inactivity will diminish the exercise improved fat metabolism after meal.

12 male and female participants will be recruited from Austin community to participate this study. All participants will self-report that they have been medically cleared for exercise by submitting a health history questionnaire. Researchers will screen all forms filled out by participants and confirm that participants are eligible for this study. Participants will receive both written and verbal descriptions of the study procedures and measurements, and provide written informed consent.

The study requires at least 7 visits besides the day for questionnaire filling and informed consent signing. One for incremental exercise test, and 6 for the three trials (one cycling session and one high fat tolerance tests for each trial). All visits will take place in the Human Performance Lab at the University of Texas at Austin. All participants will complete the incremental exercise test on a stationary bike (cycle ergometer) before three intervention trials in a randomized order.

During the incremental exercise test, participant will cycling on a cycle ergometer with a mask. Participant's breathing air will go through the tubes connecting with the mask. By analyzing the exhaled gas during the test, the maximal oxygen consumption (VO2max) will be measured for determining the cycling intensity for the cycling in the three trials. Between trials, there will be a washout period of at least five days. The three trials varies in length of physical inactive (4 hours, 8 hours, and 12 hours) during the day. Thus, the three trials are marked as 4-hr trial, 8-hr trial, and 12-hr trial. During the cycling sessions, participant will cycle for 1 hour at an intensity of 60-65% of VO2max (moderate intensity) on a cycling ergometer. The high fat tolerance test (HFTT) day will be the day for collecting primary data.

To highlight the effect of physical inactivity duration on causing exercise resistance, all HFTT will start at the same time on the testing day of each trial, which is 9 am on the final day of each trial. For easier understanding, the events sequence in each of the trails is listed below,

* One day for participant's routine steps counts and sleep hours monitor.
* A 48 hours of physical activity control phase (> 8,500 steps/24hr).
* On the third day, a physical inactivity intervention will be done either from 4 pm - 8 pm (4-hr trial), 12 pm - 8 pm (8-hour trial), or 8 am - 8 pm (12 hour trial). Hourly 600 steps will be done from the morning until the inactivity intervention starts. A 1-hr cycling session from 8 pm to 9 pm.
* A HFTT from 9 am to 2 pm on the last day of each trial.

During the whole trials, participants will be given a Fitbit wristband and a pedometer for step counts control and sleep hours record. A three day food log will be provided to participants in all trials and will be returned after each trial. A standard frozen meal will be provided to the participants to consume 2 hours before the cycling sessions to avoid the effect from fat consumption from the meal before the HFTT. Other than the sport drink that will be provided right after the cycling, participants will need to stay fasted (no food or beverage, only water) since the frozen meal to the HFTT. During the HFTT, a high fat meal (a mixture of ice cream and heavy cream) will be provided to participants. Participants will consume the milkshake in 10 min. The amount of ice cream and heavy cream will be determined by participant's body weight. During the test, five measurements (fingertip blood collection and exhaled air collection) will be done including one baseline measurement (before high fat meal), and four measurements each hour after consuming the meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between the age of 18-40 years old
* Untrained or recreationally active
* No metabolic disease, no lactose intolerance, not taking medicines altering lipid or carbohydrate metabolism
* No injury or disease affecting the cycling ability.

Exclusion Criteria:

* On medications that alter lipid or carbohydrate metabolism lactose intolerant
* General health problems: Heart problems or coronary artery disease, hypertension, lung or respiratory problems.
* Exercise problems: Chest pain, fainting, palpitations, told to give up sports because of health problems.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Fat oxidation (fat burning) | Through study completion, around 9 months
  Exhaled gas will be collected during the high fat tolerance test. Fat oxidation will be calculated based on the gas volume and CO2 and O2 proportion.
Plasma triglyceride | Through study completion, around 9 months
  Fingertip blood will be collected during the high fat tolerance test.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coyle EF, Burton HM, Satiroglu R. Inactivity Causes Resistance to Improvements in Metabolism After Exercise. Exerc Sport Sci Rev. 2022 Apr 1;50(2):81-88. doi: 10.1249/JES.0000000000000280. PMID 35025844